CLINICAL TRIAL: NCT01605383
Title: A Pilot Clinical Trial of "ex Vivo" Expanded Autologous Bone Marrow Mesenchymal Stem Cells Fixed in Allogenic Human Bone Tissue (XCEL-MT-OSTEO- ALPHA) in Osteonecrosis of the Femoral Head
Brief Title: Mesenchymal Stem Cells in Osteonecrosis of the Femoral Head
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government); Ministerio de Ciencia e Innovación, Spain (Other Government); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XCEL-MT-10-01; 2010-023998-18 (EudraCT Number)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Avascular Necrosis of Femur Head
Keywords: Avascular Necrosis of Femur Head; Osteonecrosis of the hip; Osteonecrosis of the femoral head; Mesenchymal Stem Cells; Bone marrow; Tissue engineering; Bone Diseases; Musculoskeletal Diseases
MeSH Terms: conditions — Femur Head Necrosis; Legg-Calve-Perthes Disease; Bone Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XCEL-MT-OSTEO-ALPHA (Experimental): "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue (under Xcelia-GMP conditions)for osteonecrosis of the femoral head
  Interventions: Biological: XCEL-MT-OSTEO-ALPHA
- Standard Treatment (Sham Comparator): Isolated core decompression
  Interventions: Procedure: Standard treatment

INTERVENTIONS:
Biological: XCEL-MT-OSTEO-ALPHA — Core decompression plus XCEL-MT-OSTEO-ALPHA
  Arms: XCEL-MT-OSTEO-ALPHA
Procedure: Standard treatment — Isolated core decompression
  Arms: Standard Treatment

SUMMARY:
The present study evaluates the effect of XCEL-MT-OSTEO-ALPHA in osteonecrosis of the femoral head in comparison to the standard treatment of isolated core decompression.

XCEL-MT-OSTEO-ALPHA is a tissue engineering product composed by "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue.

The working hypothesis proposes that the tissue engineering is a valid and useful technique to achieve bone regeneration, avoiding the progression to collapse of the femoral head.

DETAILED DESCRIPTION:
Prospective, open-label with blinded assessor, randomized, parallel, single-dose phase I-II clinical trial in which 24 patients affected with osteonecrosis of the femoral head ARCO grade I or II will enter the trial with the primary objective of assessing the feasibility and safety of "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue in osteonecrosis of the femoral head. Secondary objectives are to assess the efficacy of the implantation by imaging (magnetic resonance imaging) and clinical questionnaires (pain by visual analogue scale, quality of life by SF-36 and WOMAC Index).

Patients will be randomized to one of the two treatment arms (core decompression and the tissue engineering product composed by "ex-vivo" expanded autologous mesenchymal stem cells fixed in allogenic bone tissue or the standard treatment of isolated core decompression). Thereafter, patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age (male and female)
* Osteonecrosis of the hip ARCO grade I or II
* Abscence of systemic or local infection
* Laboratory tests with no relevant abnormal findings that contraindicate the surgery.
* Informed Consent Form signed
* The patient is able to understand the nature of the study

Exclusion Criteria:

* Osteonecrosis of the hip secondary to femoral neck fracture
* Patients with no closed cartilage
* Surgical implants in the femoral head
* Septic arthritis
* Patients with severe renal insufficiency
* Patients expecting or with liver transplantation
* Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg), Hepatitis C (Anti-HCV-Ab) or Syphilis.
* Pregnant woman or intended to become pregnant, or breath feeding
* Neoplasia within the previous 5 years, or without remission
* Immunosuppressive states
* The patient is legally dependent
* Participation in another clinical trial or treated with an investigational medicinal product the previous 30 days
* Cardiac pacemaker, allergy to contrast or any other condition that contraindicates the MRI with contrast agents
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria
* The patient does not accept to be followed-up for a period thar could exceed the clinical trial length

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Safety of XCEL-MT-OSTEO-ALPHA in osteonecrosis of the femoral head | 12 months
  Safety will be assessed by collecting adverse events throughout the experimental phase, which includes a follow-up of 12 months
Feasibility of XCEL-MT-OSTEO-ALPHA in osteonecrosis of the femoral head | 12 months
  Feasibility will be measured by assessing the percentage of patients to which bone marrow puncture is made are thereafter treated and by checking the cascade of procedures to confirm the global process is viable.

SECONDARY OUTCOMES:
Bone regeneration by measuring the necrotic angle using the modified Kerboul method | 6 and 12 months
  The necrotic angle will be measured using imaging procedures (magnetic resonance imaging MRI).
Dynamic changes of signal intensity | 6 and 12 months
  Dynamic changes of signal intensity after Gd enhancement in the necrotic areas of the femoral head
Clinical outcomes (pain) by Visual Analogue Scale (VAS) | 7 days and at 3, 6 and 12 months
  Pain measurement by VAS
Clinical outcomes (SF-36) | 3, 6 and 12 months
  This clinical outcome will measure the quality of life by the self-reported quality of life questionnaire SF-36
Clinical outcome (WOMAC) | 3, 6 and 12 months
  To assess the extent by which a person's functional level is restricted by the WOMAC index

CONTACTS AND LOCATIONS:
Overall Officials: Màrius Aguirre, MD, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Derived] Vives J, Oliver-Vila I, Pla A. Quality compliance in the shift from cell transplantation to cell therapy in non-pharma environments. Cytotherapy. 2015 Aug;17(8):1009-14. doi: 10.1016/j.jcyt.2015.02.002. Epub 2015 Mar 10. PMID 25769789
- See also: Banc de Sang i Teixits. Xcelia-División de Terapias Avanzadas. — http://www.bancsang.net/
- See also: Hospital Universitari Vall d'Hebron, Barcelona — http://www.vhebron.net/